CLINICAL TRIAL: NCT06999707
Title: Photon Radiotherapy Combined With Tremelimumab and Durvalumab for BCLC Stage B and C Hepatocellular Carcinoma
Brief Title: Photon Radiotherapy Plus Tremelimumab/Durvalumab for BCLC Stage B and C HCC
Acronym: Photon-STRIDE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202500671A3
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: HCC - Hepatocellular Carcinoma; Tremelimumab; Durvalumab; Radiotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tremelimumab; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Photon radiotherapy combined with Tremelimumab and Durvalumab (Experimental): Patients undergo photon radiotherapy combined with Tremelimumab and Durvalumab.
  Interventions: Radiation: Photon radiotherapy; Drug: Tremelimumab; Drug: Durvalumab

INTERVENTIONS:
Radiation: Photon radiotherapy — * 39.6-72.6 Gy in 22 fractions for tumors ≤1 cm from hepatic hilum, bowel, and heart.
  * 30-66 Gy in 10 fractions for tumors >1 cm from hepatic hilum, bowel, and heart.
  * 27.5-50 Gy in 5 fractions using stereotactic body radiation therapy (SBRT) techniques
Drug: Tremelimumab — Tremelimumab 300 mg will be administered as an IV infusion for one dose
Drug: Durvalumab — Treatment Duration Guidelines: * Complete Response (CR): Patients who achieve a CR within one year of treatment will continue durvalumab for a total duration of two years. * Partial Response (PR): Patients who achieve a PR should continue durvalumab until achieving CR, disease progression (PD), or for a total duration of two years. * Stable Disease (SD): Patients with SD will receive duvalumab for a total of 6 doses.

SUMMARY:
Tremelimumab plus durvalumab (the STRIDE regimen) is an approved first-line therapy for unresectable hepatocellular carcinoma (HCC); however, it demonstrates limited efficacy, with an objective response rate (ORR) of only 20.1%. Radiation therapy (RT) is highly effective in controlling localized solid tumors and has become an integral component of the treatment algorithm for unresectable HCC. Preclinical studies have shown that combining RT with PD-L1/PD-1 blockade promotes immunogenic cell death and enhances antigen presentation by dendritic cells, thereby boosting systemic T cell-mediated antitumor responses in mouse models. The addition of CTLA-4 inhibition further enhances antigen cross-priming following RT. Recent retrospective data also indicate that combining RT with immune-oncology agents is associated with improved overall survival and prolonged time to progression compared to RT or immunotherapy alone. However, the clinical benefit and immunologic impact of combining RT with tremelimumab and durvalumab have not yet been evaluated in prospective clinical trials for unresectable HCC.

This phase II, single-arm clinical trial aims to assess the safety, efficacy, and immunologic effects of combining proton RT with tremelimumab and durvalumab in patients with unresectable HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have diagnosis of HCC that is deemed unsuitable for surgical resection or transplant. Participants may have multiple lesions with a total maximal tumor dimension of < 20 cm, and no one lesion > 15 cm. Diagnosis should be confirmed by at least 1 criterion listed below:

   * Histologically or cytologically proven diagnosis of HCC.
   * Typical arterial enhancement and delayed washout on multiphasic CT or MRI.
2. Age ≥18 years at the time of signing informed consent document.
3. ECOG performance status 0-1.
4. Barcelona Clinic Liver Cancer (BCLC) stages Intermediate (B) or Advanced (C).
5. Child-Pugh score 5-6 liver function within 28 days of study registration.
6. Documented virology status of hepatitis B virus (HBV), as confirmed by screening HBV serology test.
7. Documented virology status of hepatitis C virus (HCV), as confirmed by screening HCV serology test.
8. Ability to understand and the willingness to sign a written informed consent document
9. Adequate bone marrow, liver, and renal function within 4 weeks before study registration

   * Hemoglobin ≥ 9.0 g/dL
   * Absolute neutrophil count (ANC) ≥ 1,000/mm3
   * Platelet count ≥ 50,000/μL
   * Total bilirubin < 2.5 mg/dL
   * Serum albumin >2.8 g/dL
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × upper limit of normal (ULN)
   * Prothrombin time ≤ 6 seconds prolonged
   * Serum creatinine ≤ 1.5 mg/dL

Exclusion Criteria:

1. Prior invasive malignancy unless disease free for a minimum of 2 years
2. Prior radiotherapy to the region of the liver that would result in overlap of radiation therapy fields
3. Prior selective internal radiotherapy/hepatic arterial yttrium therapy, at any time
4. Untreated active hepatitis B or hepatitis C
5. Moderate to severe or intractable ascites
6. Presence of distant metastases that cannot be encompassed by photon radiotherapy
7. Untreated or incomplete treated esophageal or gastric varices
8. Severe, active co-morbidity, defined as follows:

   * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months prior to registration
   * Myocardial infarction within the last 6 months prior to study entry
   * Acute bacterial or fungal infection requiring intravenous antibiotics within 28 days prior to study entry
   * A bleeding episode within 6 months prior to study entry due to any cause.
   * Thrombolytic therapy within 28 days prior to study entry.
   * Known bleeding or clotting disorder.
   * Uncontrolled psychotic disorder
9. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception
10. Prior solid organ transplantation.
11. Prior or active autoimmune disease (AID) including autoimmune hepatitis, inflammatory bowel disease, myasthenia gravis, systemic lupus erythematosus, rheumatoid arthritis, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, and multiple sclerosis.
12. Inability to treat all sites of disease by photon radiotherapy (such as extrahepatic metastases or massive liver tumors whereby the liver constraints cannot be met for covering all sites of liver tumors using photon radiotherapy.)
13. Known HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2030-05-31 (Estimated); Study Completion 2033-05-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 12 months
  Progression free survival is defined as the time from signing the informed consent to the first occurrence of disease progression or death from any cause (whichever occurs first) according to RECIST1.1

SECONDARY OUTCOMES:
Local control | 12 months
  Local control is defined as the time from signing the informed consent to the first occurrence of disease progression in the irradiated field according to RECIST1.1
Time to progression | 12 months
  Time to progression is defined as the time from signing the informed consent to the first occurrence of disease progression according to RECIST1.1
Overall Response Rate | 12 months
  Overall Response Rate is defined as a complete or partial response according to RECIST1.1
Overall survival | 12 months
  Overall survival is defined as the time from signing the informed consent to death from any cause.
Incidence and severity of adverse events | 12 months
  Description: Adverse events will be graded using CTCAE v5

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital at Linkou, Taoyuan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
Sharing individual participant data (IPD) with other researchers requires IRB review and approval. Presently, we do not have a plan to provide IPD to other researchers.